CLINICAL TRIAL: NCT01954524
Title: A Phase 1, Open-Label Study of Intravenous Sildenafil in Patients With Cirrhosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is closed due to lack of funding to support the study.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00057016
Record Dates: First submitted 2013-09-13; First posted 2013-10-01 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV bolus injection of Sildenafil (Experimental): CTP class B cirrhosis: A single 5 and 10 mg IV bolus injections of Sildenafil. CTP class C cirrhosis: A single 2.5, 5, 8 and 10 mg IV bolus injections of Sildenafil.
  Interventions: Drug: IV bolus injection of Sildenafil

INTERVENTIONS:
Drug: IV bolus injection of Sildenafil — Dose escalation will be performed (in different participants). The doses will be as follows:
  CTP class B cirrhosis: A single 5 and 10 mg IV bolus injections of Sildenafil. CTP class C cirrhosis: A single 2.5, 5, 8 and 10 mg IV bolus injections of Sildenafil.
  Other Names: Revatio

SUMMARY:
Safety and tolerability of a single dose intravenous bolus injection of Sildenafil in patients with moderate to severe cirrhosis and kidney disease will be determined.

ELIGIBILITY:
Subjects will be eligible for the study if they meet the following inclusion criteria:

1. Cirrhosis. Diagnosis of cirrhosis will be based on either liver biopsy OR clinical characteristics (e.g. history of ascites or encephalopathy or esophageal varices or gastric varices or splenomegaly or spider angioma or any clinical sign of portal hypertension/cirrhosis), laboratory (e.g. history of thrombocytopenia or history of APRI (Reference: Wai CT, Greenson JK, Fontana RJ, Kalbfleisch JD, Marrero JA, Conjeevaram HS, Lok AS. A simple noninvasive index can predict both significant fibrosis and cirrhosis in patients with chronic hepatitis C. Hepatology 2003;38:518-26) [Aspartate aminotransferase (AST) to platelet ratio index] score consistent with cirrhosis or history of abnormal liver function tests) and abdominal imaging (Magnetic Resonance Imaging or Computed Tomography or ultrasound of the abdomen) data
2. CTP Class B or C cirrhosis
3. Age 18 years or older at the time of enrollment
4. Variceal screening with an upper endoscopy within 1 year before enrollment
5. Renal dysfunction [GFR ≥ 15 and < 60 ml/min/1.73m2 estimated by 6-variable MDRD equation (Reference: Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med 2006;145:247-54)]
6. Hemoglobin level ≥ 8 mg/dl within 4 weeks before enrollment
7. Serum sodium level ≥ 125 mmol/L within 4 weeks before enrollment

Subjects will be excluded if they have any of the following:

1. Inability to provide informed consent
2. Women who are pregnant, breast-feeding, or contemplating pregnancy
3. Treatment with organic nitrates, ritonavir, erythromycin, saquinavir, ketoconazole, itraconazole, cimetidine, bosentan, rifampin, Sildenafil or any other PDE-5 inhibitors, alpha-blockers, and anticoagulants within 7 days before enrollment
4. Hypersensitivity or allergy to Sildenafil or any component of Sildenafil
5. Previous reaction to PDE-5 inhibitors including, but not limited to Sildenafil, Vardenafil, Tadalafil, Avanafil (Myocardial infarction, ventricular arrhythmia, sudden cardiac death, cerebrovascular hemorrhage, transient ischemic attack, stroke, transient global amnesia, subarachnoid and intracerebral hemorrhages, seizure, recurrence in seizures, pulmonary hemorrhage, sudden decrease of hearing, loss of hearing, anxiety, prolonged erection, priapism, ocular redness, ocular burning, diplopia, temporary vision loss/decreased vision, ocular swelling, ocular pressure, increased intraocular pressure, retinal problems in the eye, vitreous detachment, vitreous traction, paramacular edema, non-arteritic anterior ischemic optic neuropathy)
6. History of untreated severe left ventricular outflow obstruction (e.g. aortic stenosis, idiopathic hypertrophic subaortic stenosis)
7. History of pulmonary veno-occlusive disease
8. History of unstable angina, myocardial infarctus, life-threatening arrhythmia or stroke within 6 months before enrollment
9. History of retinitis pigmentosa
10. Anatomical deformation of the penis (Peyronie's disease, angulation, cavernosal fibrosis)
11. History of sickle cell anemia, multiple myeloma or leukemia
12. Renal failure treated with dialysis
13. Cognitive impairment based on IRB "evaluation to sign consent form"
14. Transjugular intrahepatic porto-systemic shunt placement
15. Previous kidney or liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with "suspected adverse reaction" of IV Sildenafil that is both "serious" and "unexpected" as a measure of safety and tolerability. | The total time to assess the primary outcome measure will be 48 hours after Sildenafil injection (starting from Sildenafil injection time until 48 hours after Sildenafil injection).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Mindikoglu AL, Dowling TC, Schaub DJ, Hutson WR, Potosky DR, Christenson RH, Barth RN, LaMattina JC, Hanish SI, Weir MR, Raufman JP. Pharmacokinetics and Tolerability of Intravenous Sildenafil in Two Subjects with Child-Turcotte-Pugh Class C Cirrhosis and Renal Dysfunction. Dig Dis Sci. 2015 Nov;60(11):3491-4. doi: 10.1007/s10620-015-3771-0. Epub 2015 Jul 5. PMID 26143343